CLINICAL TRIAL: NCT00946179
Title: Immunogenicity and Safety of the Influenza Vaccine (Split Virion, Inactivated), Northern Hemisphere 2009-2010 Formulation (Intramuscular Route)
Brief Title: Study of Influenza Vaccine (Split Virion, Inactivated) Northern Hemisphere 2009-2010 Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRT86
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Split virion
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Participants aged 18 to 60 years at enrollment
  Interventions: Biological: Influenza virus (split virion, inactivated) vaccine
- Group 2 (Experimental): Participants aged 61 years or older at enrollment
  Interventions: Biological: Influenza virus (split virion, inactivated) vaccine

INTERVENTIONS:
Biological: Influenza virus (split virion, inactivated) vaccine — 0.5 mL, Intramuscular
  Other Names: Influenza Vaccine Northern Hemisphere 2009-2010 formulation

SUMMARY:
This study is in support of the annual application for the variation of the vaccine strains for a marketing authorization.

Objectives:

* To evaluate the compliance, in terms of immunogenicity, of the influenza vaccine (split virion, inactivated) Northern Hemisphere (NH) 2009-2010 formulation in two adult groups, aged 18 to 60 years and aged 61 years or older.
* To describe the safety of the influenza vaccine (split virion, inactivated) NH 2009-2010 formulation in both adult groups.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 60 years (i.e., to the day before the 61st birthday) or 61 years or older (from the day of the 61st birthday) on the day of inclusion
* Provision of a signed informed consent
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential: avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 3 weeks after vaccination

Exclusion Criteria :

* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test at Visit 1
* Febrile illness (temperature ≥ 38 °C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to eggs, chicken proteins, neomycin, formaldehyde and octoxynol-9, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 3 weeks following the trial vaccination
* Previous vaccination against influenza in the previous 6 months
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion
* Known human immunodeficiency virus (HIV), Hepatitis B surface (HBs) antigen or Hepatitis C seropositivity
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of intramuscular (IM) Influenza Vaccine (Split Virion, Inactivated), Northern Hemisphere 2009-2010 Formulation. | 21 days post-vaccination
To provide information concerning the safety of intramuscular (IM) Influenza Vaccine (Split Virion, Inactivated), Northern Hemisphere 2009-2010 Formulation | 0 to 7 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Switzerland (2):
  - Allschwil
  - Zurich

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com